CLINICAL TRIAL: NCT04563910
Title: Impact of Duration of Untreated Bipolar Disorder (Manic Episodes) on Clinical Outcome
Brief Title: Impact of Duration of Untreated Manic Episodes on Clinical Outcome
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maggi Raoof, Maggi Raoof Samaan, Assiut University
Other Study IDs: 17101199
Record Dates: First submitted 2020-09-19; First posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Patients Diagnosed With Bipolar Disorder ( Manic Episodes) and Delayed Diagnosis
MeSH Terms: conditions — Mania

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- less than 2 episodes: Patients were classified into 3 groups according to number of episodes (1-2 episodes, 3-5 episodes, more than 5 episodes)
  Interventions: Other: young mania rating scale
- 2-5 episodes: Patients were classified into 3 groups according to number of episodes (1-2 episodes, 3-5 episodes, more than 5 episodes)
  Interventions: Other: young mania rating scale
- more than 5 episodes: Patients were classified into 3 groups according to number of episodes (1-2 episodes, 3-5 episodes, more than 5 episodes)
  Interventions: Other: young mania rating scale

INTERVENTIONS:
Other: young mania rating scale — questionnaires to the patients and their family after their written consent
  Other Names: socioeconomic scale

SUMMARY:
The current study is cross sectional retrospective study, included 100 patients were diagnosed as mood disorder bipolar I (manic episodes) according to DSM5, patients recruited from inpatient psychiatric unit at department of Neurology and Psychiatry, Assiut University hospitals The current work is designed to study the effect of duration of untreated bipolar disorder on clinical outcome ( severity , residual symptoms ,duration of hospital admission) and to study factors affecting duration of untreatment in Upper Egypt.

DETAILED DESCRIPTION:
Mood disorder carries a major burden in our country as it represents 15% of inpatients and 20% of outpatients in mental hospitals in Egypt

The current work is designed to study the effect of duration of untreated bipolar disorder on clinical outcome ( severity , residual symptoms ,duration of hospital admission) and to study factors affecting duration of untreatment in Upper Egypt.

The current study is cross sectional retrospective study, included 100 patients were diagnosed as mood disorder bipolar I (manic episodes) according to DSM5, patients recruited from inpatient psychiatric unit at department of Neurology and Psychiatry, Assiut University hospitals

ELIGIBILITY:
Inclusion Criteria:

* -Age group between 18 to 45 years old.
* Patients diagnosed as mood disorder bipolar I manic episode according to DSM V(2).
* Clearly consenting to participate in the study.

Exclusion Criteria:

* -Mood disorder due to substance abuse.
* Patients in depressive episodes.
* other mental disorders

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 patients recruited from inpatient psychiatric unit at department of neurology and psychiatry, Assiut University Hospitals
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-23 (Estimated); Primary Completion 2021-09-23 (Estimated); Study Completion 2021-10-24 (Estimated)

PRIMARY OUTCOMES:
measure the effect of duration of untreated bipolar disorder on severity (young mania rating scale on admission | one year
  To study the effect of duration of untreated bipolar disorder (manic episodes) on clinical outcomes (severity).

SECONDARY OUTCOMES:
To measure the effect of duration of untreated bipolar disorder (manic episodes) on clinical outcomes (severity, residual symptoms, duration of admission). | one year
  residual symptoms measured by young mania rating scale on discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
i will share after finishing my research

REFERENCES:
- See also: Related Info — https://www.scielo.br/scielo.php?pid=S1516-44462016005016104&script=sci_arttext